CLINICAL TRIAL: NCT06736782
Title: Holistic Self-Empowerment Care Intervention for Optimized Independent Living and Quality of Life: A Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Christian Family Service Centre (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA240023
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Long-Term Care; Caregiver Burden
Keywords: Self-Empowerment; Caregiving; Long-term Care; Hong Kong
MeSH Terms: conditions — Caregiver Burden | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A multi-site quasi-experimental study is planned to evaluate the feasibility, acceptability, and effectiveness of a Self-Empowerment Care model tailored for frail older adults in Hong Kong. Participants will be allocated into one intervention group and one control group, with the intervention group receiving a 12-week program focused on hydration, exercise, dietary support, and defecation care. This model, rooted in Nordic re-enablement principles and adapted in Japan, aims to enhance participants' independence in activities of daily living (ADLs) and quality of life (QOL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Empowerment Care Intervention Group (Experimental): Participants in the experimental group will receive a 12-week intervention based on the Self-Empowerment Care model.
  Interventions: Behavioral: Self-Empowerment Care Intervention Group
- Control Group (Active Comparator): Participants in the control group will receive usual care provided in their respective care settings. This includes routine assistance with daily activities, basic medical support, and general health monitoring without the structured interventions specific to the Self-Empowerment Care model.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Self-Empowerment Care Intervention Group — The intervention emphasizes four key principles: hydration, exercise, dietary support, and defecation care. Each component is designed to address fundamental needs and promote independence in activities of daily living (ADLs).
  Individualized care plans will be developed in collaboration with healthcare professionals and caregivers to ensure alignment with participants' functional capabilities and personal goals.
  Arms: Self-Empowerment Care Intervention Group
Behavioral: Control Group — Standard caregiving practices without emphasis on structured hydration, exercise, or dietary programs.
  General assistance with ADLs as per existing care routines in the respective facilities.
  Arms: Control Group

SUMMARY:
This protocol describes a pilot study evaluating the effectiveness of the Self-Empowerment Care Model in promoting independence and quality of life among frail older adults in Hong Kong. Rooted in Nordic re-enablement principles and refined in Japan, the intervention adopts a holistic approach that focuses on hydration, exercise, diet, and defecation care. This 12-week intervention will be tested across three care settings-residential, day care, and home care. The study uses a quasi-experimental design involving 60 participants, aiming to compare outcomes of the intervention group with a control group receiving standard care. The study also assesses its impact on caregivers' burden and job satisfaction.

DETAILED DESCRIPTION:
Introduction:

As populations age, maintaining independence in activities of daily living (ADLs) becomes essential to enhance quality of life (QOL) and reduce caregiver burden. However, traditional custodial practices often exacerbate functional decline among older adults. The Self-Empowerment Care model emphasizes enhancing independence through tailored interventions addressing physical, social, and cultural needs. Despite its successful implementation in Japan and Taiwan, its application in Hong Kong remains unexplored.

Objectives:

Evaluate the feasibility, acceptability, and effectiveness of the Self-Empowerment Care model in improving ADLs and QOL for frail older adults.

Assess the impact on caregivers, including reduced burden and enhanced job satisfaction.

Identify factors affecting the sustainability of the intervention.

Methods:

Study Design: Quasi-experimental with a 1:1 allocation ratio.

Participants:

Older adults aged ≥65 years with functional decline. Informal and formal caregivers participating voluntarily. Exclusion: severe cognitive or mental illness, terminal illness. Sample Size: 60 older adults (30 per group), plus caregivers.

Intervention: Four components:

* Hydration: Promote daily water intake of 2000 mL.
* Exercise: Sequential activities tailored by physiotherapists.
* Defecation Care: Personalized interventions based on habits.
* Dietary Support: Nutritionally balanced meals and independent eating. Control Group: Standard care without structured interventions.

Data Collection:

Quantitative: ADLs (Barthel Index), QOL (EQ-5D-5L), caregiver burden (Zarit Interview), and caregiver satisfaction (Minnesota Satisfaction Questionnaire).

Qualitative: Focus groups with caregivers to explore their experiences. Timeline: Pre- and post-intervention assessments with a follow-up focus group. Analysis A mixed-method approach will be used. Quantitative data will undergo statistical analyses (e.g., linear mixed-effects models) to compare outcomes between intervention and control groups. Qualitative data will be analyzed thematically.

Ethics and Dissemination:

Approved by the Human Research Ethics Committee of the University of Hong Kong, the study prioritizes participants' dignity and autonomy. Results will be disseminated through academic publications and shared with policymakers to inform eldercare practices.

Significance:

This study is among the first in Hong Kong to implement and evaluate the Self-Empowerment Care model. It aims to provide empirical evidence for integrating holistic eldercare models into routine practices, with the potential to benefit both aging individuals and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Functional decline
* Potential to benefit from reablement.

Exclusion Criteria:

* Severe cognitive impairment, those with mild impairment will be considered.
* Severe mental illness
* Terminal illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | 12 Weeks
  Evaluates participants' ability to perform basic activities of daily living (ADLs) independently. Scores range from 0 to 100, with higher scores indicating greater independence.
EQ-5D-5L | 12 Weeks
  A standardized instrument measuring health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Adult Social Care Outcomes Toolkit (ASCOT) | 12 Weeks
  Assesses quality of life in the context of social care, with higher scores indicating better social care outcomes.
Self-Determination Survey | 12 Weeks
  Measures participants' autonomy and motivation in managing their own care, capturing changes in self-determination over time.
Instrumental Activities of Daily Living (IADL) | 12 Weeks
  Evaluates participants' ability to perform more complex daily tasks, such as managing finances and medication, with higher scores reflecting better functionality.

SECONDARY OUTCOMES:
Minnesota Satisfaction Questionnaire (MSQ) | 12 Weeks
  Measures job satisfaction among formal caregivers, with higher scores indicating greater satisfaction in their caregiving roles.
Zarit Caregiver Burden Interview (ZBI) | 12 Weeks
  Evaluates the emotional, physical, and financial burden experienced by informal caregivers, with higher scores indicating greater burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Sau Po Centre on Ageing, HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No